CLINICAL TRIAL: NCT02995473
Title: Multi-center, Randomized, Vehicle-controlled, Investigator-blinded, Parallel Groups Study to Evaluate the Efficacy and Safety of NP000888 in Subjects With Plaque and Nail Psoriasis
Brief Title: Efficacy and Safety Study of NP000888 in Subjects With Plaque and Nail Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.100535
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NP000888 (Experimental): Pharmaceutical form: Ointment
  Interventions: Drug: NP000888
- Vehicle (Placebo Comparator): Pharmaceutical form: Ointment
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: NP000888 — 270 µg/g topical (BID) for 24 weeks
  Arms: NP000888
Drug: Vehicle — Topical (BID) for 24 weeks
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
This study is to evaluate the efficacy and safety of topical application of NP000888 ointment compared to vehicle in plaque and fingernail psoriasis subjects.

Duration of administration: 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Subject with a clinical diagnosis of plaque psoriasis defined as an IGA score at least 2 (mild) at Screening and Baseline visits
* Subject with a plaque psoriasis total Body Surface Area (BSA) involvement of at least equal to 3% but less than 20% at Screening and Baseline visits
* Subject with a clinical diagnosis of fingernail psoriasis on at least 1 fingernail with a fingernail PGA score from 2 (mild) to 4 (severe) at Screening and Baseline visits

Exclusion Criteria:

* Subject with guttata, erythrodermic, exfoliative, inverse, pustular or palmo plantar, infected or ulcerated psoriasis or psoriasis involvement >=20% BSA or an unstable form of psoriasis, defined as at least one flare in the previous month before Screening visit
* Subject with chronic plaque psoriasis who are candidates for systemic therapy at Screening and Baseline visits
* Subject with clinical signs of psoriatic arthritis at Screening and Baseline visits
* Subject with a clinical diagnosis of fingernail psoriasis on at least 1 fingernail with a nail-PGA score from 2 (mild) to 4 (severe) at Screening and Baseline visits.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Success rate in IGA score (clear or almost clear) | Baseline - Week 12
  Success rate in IGA score (clear or almost clear)
Percent change from baseline in total mtNAPSI scores | Baseline - Week 24
  Mean percent change from baseline in total mtNAPSI scores

CONTACTS AND LOCATIONS:
Locations (10):
- Taiwan (10):
  - Galderma Investigational Site, Lincuo, Taoyuan
  - Galderma investigational site, New Taipei City
  - Galderma investigational site, Taichung
  - Galderma investigational site, Tainan
  - Galderma investigational site 1, Taipei
  - Galderma investigational site 2, Taipei
  - Galderma investigational site 3, Taipei
  - Galderma investigational site 4, Taipei
  - Galderma investigational site 5, Taipei
  - Galderma investigational site 6, Taipei

IPD SHARING:
Plan to Share IPD: No